CLINICAL TRIAL: NCT06830343
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetic of SYH9017 in Chinese Participants With Overweight and Obesity Following Single and Multiple Doses
Brief Title: The Safety, Tolerability, and Pharmacokinetics of of SYH9017 in Chinese Participants With Overweight and Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH9017-001
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Overweight or Obesity
Keywords: overweight or obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SYH9017 SAD experimental group (Experimental): Subjects in SAD experimental groups will receive a single subcutaneous injection of SYH9017 on Day 1
  Interventions: Drug: SYH9017
- Placebo SAD group (Placebo Comparator): Subjects in SAD placebo groups will receive a single subcutaneous injection of placebo on Day 1
  Interventions: Drug: Placebo
- SYH9017 MAD experimental group (Experimental): Subjects in MAD experimental groups will receive subcutaneous injection of SYH9017 every 4weeks
  Interventions: Drug: SYH9017
- Placebo MAD group (Placebo Comparator): Subjects in MAD placebo groups will receive subcutaneous injection of placebo every 4weeks
  Interventions: Drug: Placebo
- Positive Control MAD group (Active Comparator): Subjects in MAD active comparator groups will receive subcutaneous injection of placebo every weeks
  Interventions: Drug: Wegovy ®

INTERVENTIONS:
Drug: SYH9017 — subcutaneous injection once time in SAD and four times in MAD
  Arms: SYH9017 MAD experimental group; SYH9017 SAD experimental group
Drug: Placebo — subcutaneous injection once time in SAD and four times in MAD
  Arms: Placebo MAD group; Placebo SAD group
Drug: Wegovy ® — subcutaneous injection once a week
  Arms: Positive Control MAD group

SUMMARY:
This is a randomized, double-blind, single-center, dose-escalation, single ascending dose and multiple ascending dose study of SYH9017 in Chinese participants with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female adult participants aged 18-60 years (inclusive) with overweight or obesity, with no less than one-third of the participants of either gender;
2. SAD phase: Body Mass Index (BMI) = weight (kg)/height^2 , with BMI in the range of 24.0-28.0 kg/m^2 (inclusive); MAD phase: Weight ≥70 kg (for males) or ≥60 kg (for females), and BMI = weight (kg)/height^2 , with BMI ≥28.0 kg/m^2;
3. Weight change <5% in the 3 months prior to screening (can be based on self-report); calculated as: (weight 12 weeks before screening - weight at screening) / weight at screening * 100%;
4. Vital signs, physical examination, 12-lead electrocardiogram, chest X-ray (anteroposterior view), abdominal color Doppler ultrasound, clinical laboratory tests (complete blood count, urinalysis, blood biochemistry, glycated hemoglobin, coagulation function, infectious disease screening, thyroid function, calcitonin, etc.) show normal results or abnormal results deemed not clinically significant by the investigator;
5. Able to read and understand the written informed consent related to the study information, fully aware of the study content, process, and possible adverse reactions, voluntarily sign the informed consent form before the trial, and ensure that they will personally participate in any procedures; Participants and their partners agree to use effective non-hormonal contraception methods (such as condoms, inert intrauterine devices, female barrier methods [cervical cap or diaphragm with spermicide], vaginal contraceptive rings, etc.) from the time of signing the informed consent form until 6 months after the last dose, or have already adopted permanent contraception measures (such as bilateral tubal ligation, vasectomy, etc.); Male participants do not plan to donate sperm from the time of signing the informed consent form until 6 months after the last dose, and female participants do not plan to donate eggs from the time of signing the informed consent form until 6 months after the last dose.

Exclusion Criteria:

1. A history of severe drug or food allergies, or any participant who is judged by the investigator to potentially be allergic to the investigational drug;
2. A history of significant diseases involving the pancreas, liver, kidneys, gastrointestinal tract, skin, cardiovascular system, respiratory system, hematological system, central nervous system, or other conditions that may endanger the safety of participants or affect the absorption, metabolism, or excretion of the study drug, and are deemed unsuitable for inclusion by the investigator;
3. A history of malignancy (except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix), psychiatric disorders (such as depression, schizophrenia, bipolar disorder, or a history of suicidal ideation or behavior), epilepsy, acute biliary disease, or confirmed acute or chronic pancreatitis; participants judged by the investigator to be unsuitable for participation in this clinical study;
4. Diagnosed with diabetes, thyroid dysfunction (abnormal TSH, FT3, or FT4 levels), Cushing's syndrome, polycystic ovary syndrome, a history of glucagonoma or pheochromocytoma, or other endocrine diseases that may affect glucose metabolism, or has experienced ≥2 episodes of severe hypoglycemia or recurrent symptomatic hypoglycemia;
5. A personal or family history of medullary thyroid carcinoma (MTC) or a history of multiple endocrine neoplasia type 2 (MEN2).
6. Any one of the following criteria is met:

   i. Participants with one or more abnormal vital signs: body temperature <35.5°C or >37.2°C, pulse rate <50 beats per minute or >100 beats per minute, systolic blood pressure ≥160 mmHg or <90 mmHg, diastolic blood pressure ≥100 mmHg or <60 mmHg. A single retest is allowed, and participants with abnormalities in both tests will be excluded; ii. Any of the following laboratory abnormalities: a) Fasting plasma glucose ≥7.0 mmol/L or fasting plasma glucose <3.9 mmol/L or HbA1c level >6.5%; b) AST or ALT >2 times the upper limit of normal (ULN), total bilirubin >1.5 times ULN, deemed clinically significant by the investigator; c) Estimated glomerular filtration rate (eGFR) <90 mL/min/1.73m²; d) Serum amylase or lipase >3 times ULN; e) Blood low-density lipoprotein cholesterol (LDL-C) ≥4.40 mmol/L; f) Triglycerides (TG) ≥5.65 mmol/L.
7. During the multiple-dose phase: Use of any approved or unapproved drugs or products that may affect body weight within 6 months prior to screening, including but not limited to orlistat, phentermine-topiramate, naltrexone-bupropion, systemic steroid medications (administered intravenously, orally, or intra-articularly), antidepressants (selective serotonin reuptake inhibitors (SSRIs), noradrenaline reuptake inhibitors (SNRIs), tricyclics, tetracyclics, etc.), psychotropic medications or sedative drugs (such as imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproate, valproate derivatives, lithium salts), etc.; or use of traditional Chinese medicines, health supplements, meal replacements, or antibiotic drugs or probiotic preparations that influence gut microbiota and thereby affect body weight; or having undergone bariatric surgery within 6 months prior to screening;
8. Use of glucagon-like peptide-1 (GLP-1) receptor agonists, GLP-1 analogs (such as liraglutide, dulaglutide, lixisenatide, exenatide, albiglutide, benraliptide, polyethylene glycol loxenatide, etc.) or any dipeptidyl peptidase-4 (DPP-4) inhibitors or glucose-dependent insulinotropic polypeptide (GIP) receptor agonists within 6 months prior to signing the informed consent form.
9. Use of any prescription medications, over-the-counter medications, traditional Chinese patent medicines, herbal remedies, vitamin dietary supplements, or health products within 4 weeks prior to signing the informed consent form;
10. Habitual intake of or consumption of excessive amounts of xanthine or caffeine-containing foods, beverages, or other substances that may affect drug absorption, distribution, metabolism, or excretion within 1 month prior to screening or within 72 hours before using the investigational drug. Examples include: coffee (more than 1100 mL per day), tea (more than 2200 mL per day), cola (more than 2200 mL per day), energy drinks (more than 1100 mL per day), chocolate (more than 510 g per day);
11. Undergone surgery (including cosmetic, dental, and oral surgeries) within 6 months prior to screening or planned during the trial period, or plans to engage in vigorous physical activity (including contact sports or collision sports) during the trial period;
12. A history of drug abuse or a positive drug screening test within 1 year prior to signing the informed consent form;
13. Loss of blood or donation of more than 400 mL of blood within 3 months prior to signing the informed consent form, or receipt of blood transfusions or use of blood products;
14. Consumption of more than 14 units of alcohol per week (1 unit = 285 mL of beer; 25 mL of spirits; 150 mL of wine) within 3 months prior to signing the informed consent form, or consumption of any alcohol-containing products within 48 hours before using the investigational drug; positive baseline alcohol test (>0 mg/100 mL) or inability to abstain from alcohol during the trial period;
15. Smoking ≥5 cigarettes daily within 6 months prior to signing the informed consent form, smoking within 48 hours before using the investigational drug, or inability to cease the use of any tobacco products during the trial period;
16. Participation in any clinical trial involving investigational drugs or medical devices within 3 months prior to signing the informed consent form;
17. Pregnant and/or breastfeeding women, or women of childbearing potential with a positive pregnancy test at screening and before dosing;
18. A history of vasovagal syncope or hemophobia, or difficulty with venipuncture for any reason, making it intolerable;
19. Difficulty with subcutaneous injection administration;
20. Any other factors deemed by the investigator to make the participant unsuitable for participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs following single-dose administration of SYH9017 Description: | up to 49 days after the dosing
Incidence of AEs following multiple doses administration of SYH9017AEs of SYH 9017 following multiple doses | up to 140 days after the last dosing

SECONDARY OUTCOMES:
The Cmax of SYH9017 following single-dose | up to 49 days after the dosing
The AUC of SYH9017 following single-dose | up to 49 days after the dosing
The Tmax of SYH9017 following single-dose | up to 49 days after the dosing
The t1/2 of SYH9017 following single-dose | up to 49 days after the dosing
The CL/F of SYH9017 following single-dose | *Time Frame:up to 49 days after the dosing
The Vz/F of SYH9017 following single-dose | up to 49 days after the dosing
The proportion of patients (%) who developed binding antibodies and neutralizing antibodies following single-dose administration of SYH9017 | up to 49 days after the dosing
The percentage change in body weight from baseline of SYH9017 following single-dose | up to 49 days after the dosing
The percentage change in waist circumference from baseline of SYH9017 following single-dose | up to 49 days after the dosing
The Cmax of SYH9017 following multiple doses | up to 140 days after the last dosing
The AUC of SYH9017 following multiple doses | up to 140 days after the last dosing
The Tmax of SYH9017 following multiple doses | up to 140 days after the last dosing
The t1/2 of SYH9017 following multiple doses | up to 140 days after the last dosing
The CL/F of SYH9017 following multiple doses | up to 140 days after the last dosing
The Vz/F of SYH9017 following multiple doses | up to 140 days after the last dosing
The Cmin of SYH9017 following multiple doses | up to 140 days after the last dosing
The RAUC of SYH9017 following multiple doses | up to 140 days after the last dosing
The RCmax of SYH9017 following multiple doses | up to 140 days after the last dosing
The proportion of patients (%) who developed binding antibodies and neutralizing antibodies following multiple doses administration of SYH9017 | up to 140 days after the last dosing
The percentage change in body weight from baseline of SYH9017 following multiple doses | up to 140 days after the last dosing
The percentage change in waist circumference from baseline of SYH9017 following multiple doses | up to 140 days after the last dosing
The proportion of participants with ≥5% weight loss during the trial period of SYH9017 following multiple doses | up to 140 days after the last dosing
The proportion of participants with ≥10% weight loss during the trial period of SYH9017 following multiple doses | up to 140 days after the last dosing
The changes in body composition (including visceral, peripheral fat, and skeletal muscle) as measured by body fat analyzer after 16 weeks of treatment, compared to baseline of SYH9017 following multiple doses | up to 140 days after the last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China